CLINICAL TRIAL: NCT05827172
Title: Catheter Ablation vs. Medical Treatment in Patients With HFrEF and Persistent AF (CAEFR-AF)
Brief Title: AF Ablation for HF With Reduced EF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: Shandong University of Traditional Chinese Medicine (Other); Yuhuan Second People's Hospital (Unknown); Tongji University (Other)
Responsible Party: Principal Investigator, Xu Liu, Dr, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAEFR-AF
Record Dates: First submitted 2023-04-11; First posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Persistent Atrial Fibrillation; Heart Failure With Reduced Ejection Fraction
MeSH Terms: conditions — Atrial Fibrillation | interventions — Nutrition Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AF ablation (Experimental): The aim of the ablation procedure was to achieve isolation of all pulmonary veins and to restore sinus rhythm.Additional ablation strategies were made at the discretion of the operators.
  Interventions: Procedure: AF ablation
- Medical therapy (rate or rhythm control) (Other): The medical therapy for atrial fibrillation was administered in accordance with the guidelines that were available at the time of the trial.Efforts to maintain sinus rhythm were recommended. Among patients who were treated for rate control, the recommended criteria varied according to the age of the patient. The aim of the treatment was a ventricular rate of 60 to 80 beats. per minute at rest
  Interventions: Other: medical therapy

INTERVENTIONS:
Procedure: AF ablation — The aim of the ablation procedure was to achieve isolation of all pulmonary veins and to restore sinus rhythm.Additional ablation strategies were made at the discretion of the operators.
  Arms: AF ablation
Other: medical therapy — The medical therapy for atrial fibrillation was administered in accordance with the guidelines that were available at the time of the trial.Efforts to maintain sinus rhythm were recommended. The aim of the treatment was a ventricular rate of 60 to 80 beats per minute at rest.
  Arms: Medical therapy (rate or rhythm control)

SUMMARY:
This is an open label, multi-center, randomized parallel control clinical trial, to examining thethe clinical outcomes of AF ablation on HFrEF patients with persistent atrial fibrillation.

DETAILED DESCRIPTION:
This is an open label, multi-center, randomized parallel control clinical trial. HFrEF patients with persistent atrial fibrillation are 1:1 randomized into the AF ablation group or the medical therapy (rate or rhythm control) group. Markers of HFrEF severity, including composite of death from any cause or worsening of heart failure that led to an unplanned overnight hospitalization,exercise hemodynamics, natriuretic peptide levels, and patient symptoms. and other indicators are analyzed to demonstrate the role of AF ablation in comparing the effects of AF ablation vs usual medical therapy for HFrEF patients with persistent atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic persistent atrial fibrillation Failure or intolerance of antiarrhythmic drug therapy or unwillingness to take antiarrhythmic drugs Left Ventricular Ejection Fraction <= 40% NYHA >= II Patient is willing and able to comply with the protocol and has written informed consent Age >= 18 years Optimal therapy for HF of ≥6 weeks Suitable candidate for catheter ablation or rate control for the treatment of AF N-terminal pro-B-type natriuretic peptide (NT-proBNP)/BNP levels above predetermined levels based on prior hospitalization and baseline rhythm

Exclusion Criteria:

* LA dimension >6.0 cm Acute coronary syndrome, cardiac surgery, angioplasty or stroke within 2 months prior to enrollment Untreated hypothyroidism or hyperthyroidism Enrollment in another investigational drug or device study Woman currently pregnant or breastfeeding or not using reliable contraceptive measures during fertility age Mental or physical inability to take part in the study Severe aortic or mitral valve disease Life expectancy <1 year

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Difference in ejection fraction between groups | Time Frame: 12 months
  Difference in left ventricular ejection fraction between groups on echocardiography at 12 months

SECONDARY OUTCOMES:
Difference in NYHA class between groups | Time Frame: 12 months
Difference in BNP between groups | Time Frame: 12 months
Difference in SR survival between groups | Time Frame: 12 months
Worsening heart failure requiring unplanned hospitalization | Time Frame: 12 months
Change in 6-minute walk distance | Time Frame: 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Song Z, Wang SY, Qidong Z, Chen N, Zhang Y, Jiang W, Wu SH, Xu K, Liu Y, Liu X, Hou X, Qin M. Catheter ablation versus medical rate control for persistent atrial fibrillation in older heart failure patients with reduced ejection fraction. Heart. 2025 Aug 12;111(17):811-817. doi: 10.1136/heartjnl-2024-324668. PMID 40393692